CLINICAL TRIAL: NCT05569434
Title: 68Ga-P16-093 PET/CT Imaging in Primary and Recurrent Glioma Patients
Brief Title: 68Ga-P16-093 PET/CT Imaging in Glioma Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-GBM093
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-P16-093 and MRI scan (Experimental): Within 1 week, each patient underwent MRI scan and PET/CT scan after intravenous administration of 68Ga-P16-093, respectively.
  Interventions: Drug: 68Ga-P16-093

INTERVENTIONS:
Drug: 68Ga-P16-093 — Intravenous injection of 68Ga-P16-093 with the dosage of 1.5-1.8 MBq (0.04-0.05 mCi)/kg. Tracer doses of 68Ga-P16-093 will be used to image lesions of glioma by PET/CT.

SUMMARY:
PSMA is highly expressed on the cell surface of the microvasculature of several solid tumors, including glioma. This makes it a potentially imaging target for the detection and grading of gliomas. This pilot study was designed to evaluate the diagnostic performance of 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, which was compared with MRI in the same group of glioma patients.

DETAILED DESCRIPTION:
Glioma is the most common primary malignant brain tumor which can be divided into four grades according to different histopathological and molecular biological characteristics.Among them, glioblastoma is one of the most common types of glioma in adults (about 55%). It belongs to WHO Grade IV high-grade glioma, with a high recurrence rate, poor prognosis, and a 5-year survival rate of less than 10%. Prostate-specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. However, PSMA is also expressed by tumor cells or neovascular endothelial cells of various solid neoplasms, such as glioma. Therefore, PSMA may be an ideal target for the diagnosis of glioma. 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, with the urea fragment of a conjugate that employs the HBED-CC chelator for labeling with 68Ga(III). The HBED-based chelating ligand binds the 68Ga3+ ion with high affinity in a pseudo-octahedral N2O4 coordination sphere by its two phenolate O, two amino-acetate carboxylate O, and two amino N donor atoms. This pilot study was designed to evaluate the diagnostic performance of 68Ga-P16-093 in the same group of glioma patients, compared with MRI.

ELIGIBILITY:
Inclusion Criteria:

* glioma patients highly suggested by MRI or histologically confirmed;
* 68Ga-P16-093 PET/CT and MRI within two weeks;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | through study completion, an average of 1 year
  comparing the number of tumor detected by 68Ga-P16-093 and MRI

SECONDARY OUTCOMES:
standardized uptake value (SUV) of tumor | through study completion, an average of 1 year
  comparing the SUVmax of tumor of different grades derived from 68Ga-P16-093

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China